CLINICAL TRIAL: NCT05789693
Title: Dissemination, Implementation, and Evaluation of an Effective School-based Intervention to Promote Physical Activity in Adolescents
Brief Title: School-based Intervention to Promote Physical Activity in Adolescents in Spain: the Promoting Physical Activity in Secondary School For Health Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Hisham Bachouri-Muniesa, Principal investigator, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UZPI21/502; 622733-EPP-1-2020-1-FR-SPO-SCP (Other Grant/Funding Number: European Comission)
Record Dates: First submitted 2023-03-03; First posted 2023-03-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Activity, Motor
Keywords: Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Physical activity changes expected
  Description:
  * Develop four sessions in the Tutorial Action Plan of the school
  * Connect several subjects aligned with the messages from the tutory
  * Physical education teachers provide some insights about healty behaviours
  Interventions: Behavioral: Physical activity changes
- No intervention (No Intervention): No Physical activity changes expected
  Descrption:
  - No intervention

INTERVENTIONS:
Behavioral: Physical activity changes — Previously an initial measure (qualitative and qualitative) will be made to know the little active adolescents. At the end of the physical activity program a retention measure will be carried out to know the scope and persistence of the variables analyzed. The intervention will be developed with a frequency of three weekly sessions, of 60 minutes, in the period of the intervention, with the exception of weeks in which there is a public holiday, where there will take measures to recover the class. A schedule for the sessions will be set according to the interests of the participants and will be the same for all.
  Other Names: Promote active lifestyles; Physical activity in adolescents
  Arms: Intervention

SUMMARY:
The goal of this study is to design, adapt and implement a strategies and a teaching intervention programme to improve the adolescents physical activity in a little city of Spain, in an educational context.

Students will be divided in two groups (control and intervention) and we will apply in the intervention in one group and we will develop different strategies aimed at improve the active lifestyles in the adolescents. Researchers will compare both groups taking in to account: levels of physical activity, sedentary time, healthy diet, self-concept or different psychosocial outcomes

DETAILED DESCRIPTION:
The purpose of the project is the development of a healthy environment from educational centers. Healthy behaviors and perceptions of healthy environments of members of the educational community will be analyzed. The data processing process will be anonymous in all students. The center will receive the information corresponding to the project through the person in charge of the investigation. The center will send a letter voluntarily accepting your participation (attached) to the principal investigator (PI) of the project. The main objective of the research project presented is to improve physical activity levels in adolescents who present rates of diagnosed active impairment through the design, development and evaluation of a multilevel and multicomponent intervention program to promote healthier lifestyles. This program will follow the principles of the Socio-ecological model, teachers and parents perceptions and beliefs, with the aim of achieving greater adherence to the sports practice of adolescents.

Students of 2nd year of E.S.O would be part of this intervention program of two educational centers of a Spanish region. Through the initial measurement made to 2nd year students of E.S.O. Overall, the investigatos would expect to have a total of about 80 male and female students, with ages between 12 and 15 years. Indirectly, parents of students and teachers would also participate. In this way, identified young people who do not perform physical activity or do not reach minimum recommendable values (recommendations of World Health Organization), will be grouped in control and experimental schools.

The study variables will be:

* Qualitative data: Collected through focus groups: personal opinions about their educational center and the development of healthy environments. Estimated completion time: 45 minutes.
* Quantitative data: The data that will be required for the students in the questionnaires (students): age, gender, place of residence and data on healthy behaviors (levels of physical activity, hours of sleep, food, hours spent on screen, substance use). and influences for a healthy environment and self-concept). Estimated completion time: 45 minutes.

The focus groups and the questionnaires will be applied once the approval of the Ethical Commitee of the region has been obtained for the application of the project. Once obtained, the following day the informed consent will be provided to the families, it will be collected in 7 days and the following week the initial questionnaires will be carried out. At the end of the research in May 2022, the same questionnaires will be passed again to assess the evolution of the group in the different study variables.

Students who do not participate in the study will be invited to non-curricular activities since participation will be voluntary. When the questionnaires are completed, the center will enable a teacher "on duty" to attend to the students during the hour that the questionnaires last.

Statistical analysis: Comparisons will be made to verify that there are no differences in the baseline, using the "t" test and the χ2 test. After verifying the assumptions of normality and homoscedasticity, an analysis of covariance with three repeated measures (ANCOVA) will be performed on the outcome variables, by intention to treat (ITT), using the last observation carried forward (LOCF) method. Age, sex, and baseline scores will be included as covariates to examine differences between groups, eliminating their possible influence. The effect size will be calculated using the partial eta square value (η2). Values ≤ 0.01 correspond to a small effect size, = 0.06 with a medium size, and ≥ 0.14 with a large size. Contrasts will be made between the pretest and posttest measurements, using the corresponding "t" test. The significance level adopted will be α< 0.05.

Limitations of the study: It is a study with a reduced sample that does not want to be representative, only to see the evaluation of the variables in that context during a specific time to help the centers make decisions about their health promoting school project.The benefits of this project would be framed in different levels. In the first place, the main benefit would be obtained by the direct recipients of the project, that is, the adolescents who would see their physical activity levels increased with the positive consequences that this entails and with the development of healthier living habits. Secondly, Physical Education teachers could have new methodological and motivational tools to encourage more physical activity among their students; and the parents of these, could value the importance of physical activity and lead an active lifestyle, collaborating from the family environment to promote the objectives of this project.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Not participating in a weight loss programme
* Provide informed consent by parents, mothers or legal guardians
* Participants must be capable and willing to provide consent
* Participants must attend at least 80% of the sessions.

Exclusion Criteria:

* Unwillingness to either complete the study requirements or to be randomized into control or training group.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Physical activity and sedentary time (objectively) | 4 months
  ActiGraph accelerometer
Physical activity and sedentary time (subjectively) | 4 months
  Questionnaire: Youth Activity Profile - Spain Likert scale (worst score) 0-4 (best score)
Future intention to practice physical activity | 4 months
  Questionnaire: Ad-hoc questions about Theory of Planned Behaviour Likert scale (worst score) 1-7 (best score)

SECONDARY OUTCOMES:
Healthy and unhealthy nutrition | 4 months
  Questionnaire: Health Behavior in School Children Survey Likert scale (worst score) 0-4 (best score)
Self-concept | 4 months
  Questionnaire: Self-concept form 5 Likert scale (worst score) 1-10 (best score)
Motivation to do exercise | 4 months
  Questionnaire: Behavioral Regulation in Exercise Questionnaire - 3 Likert scale (worst score) 0-4 (best score)

CONTACTS AND LOCATIONS:
Locations (1):
- Hisham, Huesca, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to publish several research papers related to this intervention